CLINICAL TRIAL: NCT01065753
Title: Study of Wight Reduction by Life-style Modification
Brief Title: Multi-faceted Evaluations Following Weight Reduction in Subjects With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Wayne Huey-Herng Sheu, Taichung Veterans General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C07220
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2009-12

CONDITIONS: Metabolic Syndrome
Keywords: Rho kinase; Brain-derived neurotrophic factor
MeSH Terms: conditions — Metabolic Syndrome; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Life-style modification (Experimental): Life-style modification for 40 study subjects with metabolic syndrome in comparison to 25 non-obesity subjects for control.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Diet control with exercise

SUMMARY:
Central obesity, core of metabolic syndrome, has been recognized as one of the rooting factors for development of diabetes and cardiovascular disease. Although efforts have been devoted to the studies of central obesity and/or metabolic syndrome, much remained unknown as to how obesity influences cellular as well as cardiac functions, what is the central regulation of one's body weight.

Weight loss is an undisputed way to improve cardiovascular and metabolic disorders in obese individuals. Previous studies have demonstrated that weight loss by 5% of initial weight universally provide substantial benefits in these subjects. However, there are little integrated research teams, composed of different disciplines, share common weight reduction program to look at different aspects of weight reduction in non-diabetic individuals with metabolic syndrome. The significances of this proposal we plan to target, namely Rho kinase activity from peripheral leukocyte, several cardiac functions measured by noninvasive technique (VP-2000) and MRI, circulating brain-derived neurotrophic factors (BDNF) levels, are fully explained detailed in each sub-proposal.

In order to accomplish this integrated proposal, we will form research teams including endocrinologists, cardiologists, radiologists, and a coordinating data center. We pan to recruit 40 non-diabetic individuals with metabolic syndrome to participate this 12-16 weeks weight reduction program. Twenty-five age, sex matched non-diabetes lean will be served as controls. Oral glucose tolerance test, fasting blood obtained, noninvasive vascular and MRI examinations will be applied before and after weight reduction program in those achieving at least 5% loss of initial weight.

In summary, this study will investigate the effects of weight loss on (1) Rho kinase activity obtained from peripheral leukocyte; (2). Aortic stiffness, central aortic pressure and hemodynamic by a noninvasive vascular profiling system (VP-2000); (3) Brain function specifically reflecting by circulating BDNF; (4). Aortic elastic properties and left ventricular function by using MRI examinations, in non-diabetic individuals of metabolic syndrome.

DETAILED DESCRIPTION:
Obesity, in particular central obesity, has been one of the important documented risk factors for development of diabetes and cardiovascular disease. Recent re-delineated various versions of definitions of metabolic syndrome, has fueled further the critical involvement of central adiposity in these disorders through several facets, including many increased circulating pro-inflammatory cytokines, directly or indirectly linking to visceral adipose tissue expressions. Although lots of efforts have been devoted to the studies of central obesity and/or metabolic syndrome, much remained unknown as to how obesity affect cellular as well as cardiac function, what is the central regulation of one's body weight, and how to measure fat in visceral organs precisely.

Weight loss is an undisputed way to improve cardiovascular and metabolic disorders. Both a recent review article and data from us demonstrated that only weight loss by 5% of initial weight universally delivered benefits on obese individuals. However, there is little integrated research teams from different disciplines share common weight reduction protocol and look at different aspects of weight reduction in non-diabetic individuals with metabolic syndrome. The significances of this proposal we plan to target are explained in detail in each sub-proposal. However, we would like to make a briefing description here.

1. . Rho kinase (ROCK) is a serine/threonine kinase that mediates the downstream signaling of the small guanosine triphosphate- binding protein, Rho, on the actin cytoskeleton. In mostly animal models, the inhibition of ROCK ameliorates many cardiovascular conditions, including hypertension, atherosclerosis, myocardial fibrosis, and stroke. Recent study from Taiwan showed that ROCK activity is increased in patients with metabolic syndrome.
2. . Obese and overweight individuals have increased levels of arterial stiffness which is a measure of aortic and large vessel distensibility or compliance. Weight loss could induce significant reduction in sympathetic activity and blood pressure. However, little is known as whether weight loss can improve arterial stiffness, central aortic blood pressure and related hemodynamics.
3. . Brain-derived neurotrophic factor (BDNF), recently reported related to Alzheimer's disease, is present in brain tissues extensively. It is also noted that low circulating level of BDNF was associated with impaired glucose metabolism, and might be associated higher BMI or body fat. We are interesting in effect of weight reduction on circulating BDNF values in non-diabetic subjects with metabolic syndrome.
4. . Magnetic resonance imaging (MRI) of the heart is frequently used and can provide accurate and reproducible measurement of LV mass, volumes, systolic function and aortic pulse velocity. Although echo-cardiography has been applied to study effect of weight loss on cardiac function, there has been no study by using cardiac MRI to measure cine images of cardiac function and related variables before and after weight reduction in non-diabetic subjects with metabolic syndrome.

In order to accomplish this integrated proposal, we will formulate research teams including endocrinologists, cardiologists, radiologists, and a data center, coordinated by a PhD researcher (infra-structure as described below). We will recruit 40 non-diabetic individuals with metabolic syndrome (fulfilled the criteria from IDF, 2006 and DOH of Taiwan). Twenty-five age, sex matched non-diabetes lean will be served as controls.

Written informed consent will be obtained from each subject before being enrolled into the study after approval from IRB of Taichung VGH, Taichung, Taiwan. This weight reduction program will be assisted by experienced dieticians and sports experts, all of whom we had collaborated and published article previously. This program will last for 12-16 weeks with every participants join together courses 4 hours per week. Each participant will be introduced a dietary plan based on a caloric reduction of 1200 Kcal/day from the values thought necessary to maintain their usual weight. Subject will be asked to follow dietary advice and their eating habit will be reviewed by dietician at the time of their weekly visit. Activity levels will be encouraged to reach 30 min each day and at least 5 days a week. During each visit, weight of each participant will be recorded and announced. Meals replacement may considered for those did not get much improvement during weekly monitoring since recent report indicated that meals replacement may provide certain help in reducing body weight. We are confident that adequate weight reduction (at least 5% of initial weight) and good compliance will be achieved given our previous experience.

In aggregate, this study will investigate the effects of weight loss on (1) Rho kinase activity obtained from peripheral leukocyte (2). Aortic stiffness, central aortic pressure and hemodynamic by a noninvasive technique (3) Brain function specifically reflecting by circulating BDNF levels (4). Aortic elastic properties and left ventricular function by using MRI examinations, in non-diabetic individuals of metabolic syndrome. Findings from this integrated proposal will provide valuable information as mild to moderate weight loss (5% of initial body weight) in cellular, cardiac and central nervous system in additional to well-known effects on lipids, inflammatory cytokines and insulin resistance in non-diabetic subjects with metabolic syndrome.

Follow up- Subjects received physical check up, fasting blood tests and OGTT 6 and 12 months after the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* Metabolic syndrome by IDF 2005 criteria

Exclusion Criteria:

* known diabetes
* obesity due to endocrinologic disorders
* Psychological disorder or using psychological medications
* Abnormal liver function (three-fold upper normal limit)
* Abnormal renal function (1.5-fold upper normal limit)
* Investigator judgement for abnormal clinical data
* Life-threatening disease
* Acute infective status
* Alcohol or drug abuse
* pregnant potency without prevention
* receiving other clinical trial in recently three months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
change of body weight | 12-16 weeks

SECONDARY OUTCOMES:
Change of Rho kinase | 12-16 weeks
Change of central aortic blood pressure and related hemodynamics | 12-16 weeks
Change of Brain-derived neurotrophic factor | 12-16 weeks
Change of MRI images of cardiac function | 12-16 weeks
Change of profiles before and after OGTT | 12-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wayne HH Sheu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Liang KW, Tsai IC, Lee WJ, Lin SY, Lee WL, Lee IT, Fu CP, Wang JS, Sheu WH. Correlation between reduction of superior interventricular groove epicardial fat thickness and improvement of insulin resistance after weight loss in obese men. Diabetol Metab Syndr. 2014 Oct 29;6(1):115. doi: 10.1186/1758-5996-6-115. eCollection 2014. PMID 25383099
- [Derived] Lee IT, Fu CP, Lee WJ, Liang KW, Lin SY, Wan CJ, Sheu WH. Brain-derived neurotrophic factor, but not body weight, correlated with a reduction in depression scale scores in men with metabolic syndrome: a prospective weight-reduction study. Diabetol Metab Syndr. 2014 Feb 13;6(1):18. doi: 10.1186/1758-5996-6-18. PMID 24524285
- [Derived] Lee IT, Lee WJ, Tsai IC, Liang KW, Lin SY, Wan CJ, Fu CP, Sheu WH. Brain-derived neurotrophic factor not associated with metabolic syndrome but inversely correlated with vascular cell adhesion molecule-1 in men without diabetes. Clin Chim Acta. 2012 May 18;413(9-10):944-8. doi: 10.1016/j.cca.2012.02.013. Epub 2012 Feb 21. PMID 22374129